CLINICAL TRIAL: NCT03102684
Title: Clinical Impact of Secondhand Exposure to Aerosols Produced by E-cigarettes on the Respiratory System (TackSHS Project)
Brief Title: Impact of Secondhand Exposure to E-cigarettes Aerosols on the Respiratory System
Acronym: TackSHSWP6
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Hellenic Cancer Society (Other); Public Health Agency of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TackSHS WP6
Record Dates: First submitted 2017-03-03; First posted 2017-04-06 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Second Hand Tobacco Smoke
Keywords: e-cigarette; electronic cigarette; passive exposure; secondhand exposure; smoking; respiratory system
MeSH Terms: conditions — Vaping; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No exposure (No Intervention): No exposure to secondhand exposure to aerosols produced by e-cigarettes
- Low exposure (Experimental): Secondhand exposure to e-cigarette aerosols (low)
  Interventions: Other: Secondhand exposure to e-cigarette aerosols (low)
- High exposure (Experimental): Secondhand exposure to e-cigarette aerosols (high)
  Interventions: Other: Secondhand exposure to e-cigarette aerosols (high)

INTERVENTIONS:
Other: Secondhand exposure to e-cigarette aerosols (low) — Participants will be exposed to secondhand aerosols produced by e-cigarette use. E-cigarette with low resistance will be used by an experienced smoker (tobacco flavor liquid, 12 mg nicotine, 4 sec puffs, 20-30 seconds inter-puff interval). Duration of exposure: 30 minutes.
  All study subjects will participate in this arm as the study has a cross-over design.
  Arms: Low exposure
Other: Secondhand exposure to e-cigarette aerosols (high) — Participants will be exposed to secondhand aerosols produced by e-cigarette use. E-cigarette with high resistance will be used by an experienced smoker (tobacco flavor liquid, 12 mg nicotine, 4 sec puffs, 20-30 seconds inter-puff interval). Duration of exposure: 30 minutes.
  All study subjects will participate in this arm as the study has a cross-over design.
  Arms: High exposure

SUMMARY:
Limited studies have evaluated potential exposure to secondhand e-cigarette aerosol, an indication of impact on indoor air quality. Also limited are the studies regarding direct passive exposure of humans and most of these studies have limitations, such as the small number of participants, the different methodology and devices used, or the fact that they are laboratory studies, where exposure parameters differ significantly from the actual user's habit and device. Therefore, TackSHS Project has foreseen an intervention study of cross-over design in similar to real-life conditions that aims to assess the mediating effect of e-cigarette battery output on pulmonary outcomes and indexes to provide a better understanding of the extent to which passive exposure to aerosols produced by use of e-cigarette impacts exhaled NO and exhaled breath condensate metabolites.

DETAILED DESCRIPTION:
This study is a part of a larger research project (TackSHS) funded by the European Union's Horizon 2020 Research and Innovation Programme (Grant Agreement No 681040). The current study main aim is to assess the impact of passive exposure to aerosols produced by use of e-cigarettes on indexes of lung function (respiratory mechanics and exhaled biomarkers) among healthy adults.

To achieve this objective, a laboratory based intervention study of cross-over design will be conducted at the "George D Behrakis RESEARCH LAB" of the Hellenic Cancer Society. Specifically, three trial arms will be performed (no exposure to e-cigarette aerosols (1) vs. low e-cigarette aerosols exposure (2) vs. high e-cigarette aerosols exposure (3)) with each subject participating in each of the three trial arms. Each trial arm is based around two battery power outputs, one of the key factors related to the production of e-cigarette aerosols.

Sample size:

The study sample will be 40 participants. The participants will be randomized to a sequence of exposures, and thus all the participants are requested to participate in all three trial-arms. In total, 120 person-exposures will take place (3 trial-arms x 40 adults) during the duration of this study, leading to 240 pre and post measurements.

Study Population:

Recruitment will take place within a community setting in Athens (Greece) among volunteers. Two types of participants are requested:

1. Healthy non-smokers - to be exposed to e-cigarette aerosols (secondhand exposure)
2. Healthy e-cigarette users - to create the e-cigarette exposure

Intervention

An intervention for the arms 2 and 3 will be a 30-minute exposure to aerosols produced by use of e-cigarette by an experienced user. The difference between arm 2 and 3 exposure would lie in distinct opposition to electric current of the e-cigarette battery (resistance), in particularly, low (arm 2) and high (arm 3) battery resistance will be used. Each volunteer will be given appropriate information on exposure and health effects.

Measurements:

The following measurements will be performed at each arm:

* Exhaled CO
* Oscillometry
* Exhaled NO (FeNO)
* Exhaled Breath Condensate (EBC)
* Environmental measurements - PM1, PM2.5

Equipment to be used:

* Bedfont microsmokelyser
* Sidepak TSI
* Viasys, Vmax series body-box system
* Viasys, Jaeger Masterscreen IOS system: (heated pneumotach, resistance=0.05 kPa/(L/s) at 10 L/s), in line with ATS/ERS task force guidelines 2005 25
* ECO Medics, AG CLD 88 chemilluminescense, Spiroware 3.021
* Turbo-Deccs EBC
* Thermoscientific Deepfreezer

Exposures will take place within a standardized exposure chamber successfully used with similar protocols for exposure to secondhand tobacco smoke from conventional cigarettes. The chamber will allow to control for the environmental conditions of exposures and verify that the measures changes in outcomes will be attributable solely to the trial-arm.

All individuals taking part, will be informed by the responsible physician, regarding the study, the specific tests they are about to undergo, their procedure, clinical significance and impact.

The investigators will also provide answers to any possible questions, as well as information regarding the following issues:

* The purpose of the information to be collected, including aims, methods and implications of the research;
* The extent to which personal data is used and accessed by various partners (it will be made clear that all data pertaining to them is stored and handled in an anonymous manner using encrypted - not personally identifiable- codes);
* The participant's right to access personal data and/or study data; and
* The participant's right to withdraw from participation in the study, at any point, without consequences and without obligation of explanation or justification

If the individual agrees to participate, the participant will have to confirm this by reading the information sheets and providing consent to the researcher.

The results of the medical tests included in this study, will be given to all participants along with the corresponding diagnostic interpretation.

All individuals participating in this study can freely access their own personal data, but it will be made clear to the study participants that no research results from the project will be returned to the subjects. However, data related to the entire project will be publicly disseminated once it has been processed and protected. This will be accessed through the project website or through publications related to this project.

It will be made clear that the subjects are completely free to withdraw their records from participation at any time. It will be made clear that the consent given by participants in the project can be withdrawn at any time, without any explanation or justification. In this case all data pertaining to the subjects in question will be destroyed.

The results of the medical tests included in this study, will be given to all participants along with the corresponding diagnostic interpretation.

All individuals participating in this study can freely access their own personal data, but it will be made clear to the study participants that no research results from the project will be returned to the subjects. However, data related to the entire project will be publicly disseminated once it has been processed and protected. This will be accessed through the project website or through publications related to this project.

All measurements will be conducted by trained clinical researchers. Besides the information about sociodemographic characteristics, data on smoking consumption and e-cigarette use and other tobacco variables will be also collected.

Data will be saved in electronic format and protected by password. Only a selected number of pre- designated members of the data collection team will have access to these laptops. Once data collection is complete, all data will be uploaded to a single database and reliably and completely deleted from the laptops. Selected personal data, including the names of respondents, will be collected to enable quality assurance procedures and to allow participants willing to withdraw from participation in the survey to have their records deleted from the database. Once quality assurance procedures are complete (within 4 months of the completion of data collection), names and other unique personal identifiers (such as full address) will be reliably and completely deleted.

Statistical analyses will be focused on identifying both a deterministic effect as also investigation into a potential dose-response effect between lower vs. higher exposures to e-cigarette aerosols. Once the complete dataset of all participants has been merged and cleaned, the data will be analysed using SPSS.

Specific analyses will allow us to investigate the associations between exposure to e-cigarette emissions and

1. indexes of lung mechanics (impedance, resistance, reactance, resonant frequency, frequency dependence of resistance)
2. exhaled biomarkers (exhaled NO levels and EBC levels of 8-isoprostane). The model will also allow for adjustment of any potential confounding subject-level factors and will provide estimates of within and between subject variance components and correlations.

The TackSHS project is coordinated by Dr. Esteve Fernandez from Institut Catala d'Oncologia (ICO) (SPAIN). This study is managed by the "George D Behrakis RESEARCH LAB", within the Hellenic Cancer Society (HCS) (Greece), with collaboration of the Institut Catala d'Oncologia (ICO) (SPAIN) and the Public Health Agency of Barcelona (ASPB) (SPAIN) as partners.

ELIGIBILITY:
Inclusion Criteria:

For non-smokers:

* Age 18-35
* Non-smokers (exhaled CO measurement before each session), or
* Ex-smokers (> 1 year)
* Healthy as by non-significant medical history, normal physical examination and flow volume loop within predicted normal limits (ATS/ERS Task Force 2005)
* Normal BMI< 30

For e-cigarette users

* Age 18-35
* Normal BMI< 30
* Experienced e-cig users:>2 months use
* Healthy as by non-significant medical history, normal physical examination and flow volume loop within predicted normal limits (ATS/ERS Task Force 2005)

Exclusion Criteria:

For non-smokers

* Smokers of all kinds and devices, ex-smokers (< 1 year)
* Age <18, >35
* BMI>30
* Pregnancy, lactation
* Ongoing or recent illness (<4 weeks prior to study), recent infection (<4 weeks)
* Acute or chronic condition or disease (diabetes, asthma, COPD, congenital heart disease, arrhythmia, hypertension…)
* Medication of any kind (<2 weeks prior to study)

For e-cigarette users

* Non-smokers
* Age <18, >35
* BMI>30
* Pregnancy, lactation
* Ongoing or recent illness (<4 weeks prior to study), recent infection (<4 weeks).
* Acute or chronic condition or disease (diabetes, asthma, COPD, congenital heart disease, arrhythmia, hypertension…)
* Medication of any kind (<2 weeks prior to study)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Mechanical functions of respiratory system | The measurements (IOS, FeNO, EBC) will be performed in each trial arm immediately after the exposure; the 30 minutes time frame applies for the collective measurements and it is the time needed to perform all 3 tests according to the ATS/ERS guidelines.
  By means of impulse oscillometry system (IOS) the following idicators will be measured: Respiratory system total Impedance (Z5), Resistance (R5, R10, R20), Reactance (X5, X10, X20), Resonant Frequency (Rf), Frequency dependence of resistance (fdr), Area AX.
Fraction of Exhaled Nitric Oxide (FeNO) | The measurements (IOS, FeNO, EBC) will be performed in each trial arm immediately after the exposure; the 30 minutes time frame applies for the collective measurements and it is the time needed to perform all 3 tests according to the ATS/ERS guidelines.
  Measurement of airway eosinofilic inflammation

SECONDARY OUTCOMES:
Exhaled Breath Condensate (EBC) | The measurements (IOS, FeNO, EBC) will be performed in each trial arm immediately after the exposure; the 30 minutes time frame applies for the collective measurements and it is the time needed to perform all 3 tests according to the ATS/ERS guidelines.
  8 isoprostane measurement as a means for oxidative stress evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tzortzi, MD,FCCP, Principal Investigator — Hellenic Cancer Society
Locations (1):
- "George D Behrakis RESEARCH LAB" of the Hellenic Cancer Society (HCS), Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tzortzi A, Teloniatis SI, Matiampa G, Bakelas G, Vyzikidou VK, Vardavas C, Behrakis PK, Fernandez E. Passive exposure to e-cigarette emissions: Immediate respiratory effects. Tob Prev Cessat. 2018 May 7;4:18. doi: 10.18332/tpc/89977. eCollection 2018. PMID 32411845
- See also: TackSHS Project — http://tackshs.eu/